CLINICAL TRIAL: NCT05119127
Title: The Purpose of This Research is to Assess Vivity Toric IOL Rotational Stability at the End of Surgery, Post op 1 Day, Post op 1 Week and Post op 4 Weeks. Participants in This Research Study Are 45 Years of Age or Older and Have Planned Implantation in at Least One Eye With an Acrysof IQ Vivity Extended Vision Toric IOL.
Brief Title: Rotational Stability of Acrysof IQ Vivity Extended Vision Toric IOL and Refractive Visual Outcome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kevin Barber (Other)
Collaborators: Alcon Research (Industry); Eric Rosenberg, D.O.,M.Sc.Eng. (Unknown)
Responsible Party: Sponsor-Investigator, Kevin Barber, Ophthalmologist, Central Florida Eye Specialists, LLC
Organization: Central Florida Eye Specialists, LLC (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 63171943
Record Dates: First submitted 2021-11-05; First posted 2021-11-12 (Actual); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Cataract
Keywords: Vivity; Cataract; Intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: Study will include adults (45 years and older) who plan to have cataract extraction and subsequent implantation of AcrySof® IQ Vivity™Extended Vision Toric IOL in at least one eye. Approximately 40 eye will be screened to identify 35 qualified eyes. Within 40 days of screening, qualified subjects will receive cataract surgery followed by implantation of the AcrySof® IQ Vivity™Extended Vision Toric IOL at the surgery visit. If the second eye will participate in the study, subjects will receive the second eye cataract surgery within 60 days of the Screening visit 0. Four postoperative follow up visits are planned to occur at 1-2 days, 7-14 days, and 28-35 days for each enrolled eye. Subject participation in this study is expected to last up to 2 months, including a total of 5 study visits for subjects implanted in one eye and up to 9 visits for subjects implanted in both eyes. Upon completion of the 35 day follow up visit subjects will be exited from the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- vivity toric IOL implantation arm (Experimental): vivity toric intraocular lens will be implanted in one eye and undergo digital imaging intra op and post op to evaluate for toric intraocular lens rotational stability.
  Interventions: Device: Alcon Vivity toric intra ocular lens

INTERVENTIONS:
Device: Alcon Vivity toric intra ocular lens — implanting vivity toric IOL to asses rotational stability. IOL is already FDA approved for implantation at time of cataract surger. Intervention is to assess rotational stability and visual outcome.

SUMMARY:
The purpose of this research is to assess the rotational stability of the AcrySof IQ Vivity Extended Vision Toric IOL and Refractive Visual outcome.

DETAILED DESCRIPTION:
Assessment of the rotational stability and Refractive Visual Outcome of the AcrySof IQ Vivity Extended Vision Toric IOL at the end of surgery, post op 1 day, post op 1 week and post op 4 weeks. Participants in this research study are 45 years of age or older and have planned implantation in at least one eye.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing cataract extraction with intraocular lens implantation.
* Age: 45 years and older.
* Willing and able to comply with scheduled visits and other study procedures.
* Subjects who require an IOL power in the range of +15.0 D to +25.0 D.
* Subjects with regular corneal astigmatism that can be treated with T3-T5.
* Have good ocular health, with no pathology that compromises visual acuity (Outside of residual refractive error and cataract)
* Potential postoperative visual acuity of 0.2 logMAR/ETDRS (20/32 Snellen) or better in both eyes.

Exclusion Criteria:

* Glaucoma.
* Clinically significant corneal dystrophy.
* Previous corneal refractive surgery (i.e LASIK, PRK, RK)
* Pupil abnormalities.
* Concurrent infectious/non-infectious uveitis.
* History of chronic intraocular inflammation.
* Visually significant macular disease.
* History of retinal detachment.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Rotational stability of Vivity Toric IOL. | Five months
  Rotational stability of Vivity Toric IOL will be measured at post op 1 day, post op 1 week and post op 4 weeks.

SECONDARY OUTCOMES:
Percentage of eyes with residual refractive astigmatism, absolute residual astigmatism prediction error, and monocular distance and intermediate visual acuities. | Five months
  Percentage of eyes with post op rotation of five degrees or less, absolute prediction of error ≤ 0.5 D, residual astigmatism ≤ 0.5 D, residual astigmatism 1.00 D.
  Monocular and Binocular UDVA, UIVA, UNVA, CDVA, DCIVA and DCNVA.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Barber, MD, Principal Investigator — Ophthalmologist
Locations (1):
- Central Florida Eye Specialists, DeLand, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barber KM, O'Connor S, Mackinder P, Chih A, Jones B. Rotational stability and refractive outcomes of the DFT/DATx15 toric, extended depth of focus intraocular lens. Int Ophthalmol. 2023 Aug;43(8):2737-2747. doi: 10.1007/s10792-023-02673-7. Epub 2023 Mar 10. PMID 36894823